CLINICAL TRIAL: NCT00303121
Title: Compliance and Administration Technique in Topical Drug Therapy of Glaucoma
Status: Completed | Type: Observational
Sponsor: University of Toronto (Other)
Other Study IDs: UHN REB 05-0631-AE
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-06

CONDITIONS: Glaucoma
Keywords: Glaucoma; Compliance; Therapy; Administration technique
MeSH Terms: conditions — Glaucoma; Patient Compliance

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Clinic-based evaluation of patients compliance with topical medications in the treatment of glaucoma. Also assessing effectiveness of delivery techniques among these patients.

ELIGIBILITY:
Inclusion Criteria:

glaucoma 18 years of age or older

Exclusion Criteria:

Recent ocular surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-11; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne M Buys, MD, Principal Investigator — University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada